CLINICAL TRIAL: NCT05562531
Title: Evaluation of the Chewing Performance and Nutritional Status of the Patients Diagnosed With Bruxism After Botulinum Toxin Application: Follow-up Study
Brief Title: Botulinum Toxin Administration on Masticatory Performance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MU_DHF_SBF_01
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Temporomandibular Disorder; Bruxism
Keywords: Botulinum Toxins, Type A; Mastication; Nutritional Status; Bruxism; Chewing
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to evaluate the effect of botulinum toxin type A (BTX-A) injection on masticatory performance and nutritional status in temporomandibular disorder patients with bruxism caused by both intra-articular and extra-articular pathologies based on Research Diagnostic Criteria for temporomandibular disorders (TMD). The baseline and end masticatory performance, pain intensity, nutrition and anxiety statuses, and anthropometric measurements will be compared.

DETAILED DESCRIPTION:
The main purpose of this study is to determine the effect of BTX-A injection on masticatory performance and nutritional status in TMD patients with bruxism.

Sub-objectives of the study;

Determination of the effect of BTX-A on masticatory performance Determination of the effect of BTX-A on pain intensity Determination of the effect of BTX-A on anthropometric measurements Determination of the effect of BTX-A on nutritional status Determination of the effect of BTX-A on anxiety status.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years old,
* Male or female,
* Able to communicate
* Able to read and write
* Volunteer to participate in the study,
* At least 3 months of splint treatment and no results
* Having Class 1 molar occlusion and not using removable prostheses
* Marmara University, Faculty of Medicine, Department of Oral and Maxillofacial Surgery, patients diagnosed with bruxism or myofascial pain in masticatory muscles will be included in the study.

Exclusion Criteria:

* Sensitivity to botulinum toxin,
* Have received botox treatment in the last 6 months,
* Injection site infection
* Pregnant or lactating women
* Those with diseases that may cause systemic neuropathy such as diabetes, hypertension, kidney disease,
* Those who do not want to sign the consent form,
* Patients with a history of malignancy, radiotherapy or chemotherapy will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who applied to the Marmara University Faculty of Dentistry Department of Oral and Maxillofacial Surgery for bruxism and joint pain will be included in the study. It is aimed to invite all patients who applied to the clinic to the research.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the masticatory performance at 6 months | 6 months
  The masticatory performance of patients at the baseline, 1 month and 6 months later will be taken with a color-changeable gum, called "XYLITOL", (70x20x1 mm 3 g; Masticatory Performance Evaluating Gum XYLITOL, Lotte, Tokyo, Japan). Color changeable gum was first developed specifically to evaluate a person's masticatory performance; and it changes color as it is chewed. The gum will be chewed 60 times by the TMD patients. These values will be recorded and compared with the baseline, 1 month and 6 months later. After chewing, the gum colour will be evaluated according to the improved colour scale. Colour scale ranges from 1-10, and the masticatory performance will be evaluated as poor (1-6), normal (7-8), or good (9-10) with the improved color scale.
Change from baseline in the nutritional status at 6 months | 6 months
  The nutritional status of patients at the baseline, 1 month, and 6 months later will be taken with 24-hour recall method. The data obtained from the 24-hour recall method will be analyzed using the "Computer Assisted Nutrition Program, Nutrition Information Systems Package Program (BEBIS)" and the amount of energy, carbohydrates, protein, fat and fiber consumed by participants will be calculated. Intake of energy, macro nutrients and fiber will be compared with the baseline, 1 month and 6 months later.
Change from baseline in the BMI at 6 months | 6 months
  The body weight (kg) and height (m) of the patients at the baseline, and 6 months later will be taken by the researcher and noted in their files.
  The height of patients will be taken using a stadiometer with the nearest 0.1 cm, while each participant is standing erect against the wall with heels together touching the wall, without shoes.
  Body composition will be analyzed by Tanita DC-360 (Accurate Technology Co., Ltd. Tianjin, China) according to the standard procedure, and the body weight, percentage of body lean mass, and fat of the participants will be recorded. Body mass index (BMI) will be calculated using weight (in kilograms) divided by the height squared (in square meters).

SECONDARY OUTCOMES:
Change in pain intensity | 6 months
  Change in muscle pain intensity was assessed using a Visual Analogue Scale (VAS) ranging from the absence of pain (score 0) to the most severe pain imaginable. The VAS consist of a line which can be presented horizontally or vertically (10 cm long) with anchor points of "no pain" and "worst possible pain". The patient will be asked to put a mark on the line that best describe the pain severity. The patients' responses' will be recorded and scored according to the VAS scale. Than, the results will be compared with the baseline, 1 month and 6 months later.
Change from baseline in the anxiety status at 6 months | 6 months
  The anxiety status of patients at the baseline, 1 month, and 6 months later will be taken with Beck Anxiety Index. These scores will be recorded and compared with the baseline, 1 month and 6 months later.
Change in chewing ability | 6 months
  In this study, a questionnaire consisting of open and closed-ended questions will be used to determine the chewing difficulties of individuals. With open-ended questions, foods that are difficult to chew and the methods used to consume these foods will be questioned. In the follow-up interviews, closed-ended questions such as the ability to chew the previously listed foods are "easy to chew", "I have a little difficulty", "I have a lot of difficulty / can't chew at all". If individuals say, "I have a little or a lot of difficulty" while chewing hard foods and "I have some or a lot of difficulty" when chewing soft foods, they will be evaluated as "difficulty in chewing".

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Chisnoiu AM, Picos AM, Popa S, Chisnoiu PD, Lascu L, Picos A, Chisnoiu R. Factors involved in the etiology of temporomandibular disorders - a literature review. Clujul Med. 2015;88(4):473-8. doi: 10.15386/cjmed-485. Epub 2015 Nov 15. PMID 26732121
- [Background] Resende CMBM, Rocha LGDDS, Paiva RP, Cavalcanti CDS, Almeida EO, Roncalli AG, Barbosa GAS. Relationship between anxiety, quality of life, and sociodemographic characteristics and temporomandibular disorder. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Feb;129(2):125-132. doi: 10.1016/j.oooo.2019.10.007. Epub 2019 Nov 26. PMID 31784398
- [Background] Edwards DC, Bowes CC, Penlington C, Durham J. Temporomandibular disorders and dietary changes: A cross-sectional survey. J Oral Rehabil. 2021 Aug;48(8):873-879. doi: 10.1111/joor.13210. Epub 2021 Jun 11. PMID 34031904
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Haketa T, Kino K, Sugisaki M, Amemori Y, Ishikawa T, Shibuya T, Sato F, Yoshida N. Difficulty of food intake in patients with temporomandibular disorders. Int J Prosthodont. 2006 May-Jun;19(3):266-70. PMID 16752624
- [Background] Hama Y, Kanazawa M, Minakuchi S, Uchida T, Sasaki Y. Properties of a color-changeable chewing gum used to evaluate masticatory performance. J Prosthodont Res. 2014 Apr;58(2):102-6. doi: 10.1016/j.jpor.2013.12.005. Epub 2014 Jan 23. PMID 24461959
- [Background] Kamiyama M, Kanazawa M, Fujinami Y, Minakuchi S. Validity and reliability of a Self-Implementable method to evaluate masticatory performance: use of color-changeable chewing gum and a color scale. J Prosthodont Res. 2010 Jan;54(1):24-8. doi: 10.1016/j.jpor.2009.08.001. PMID 19837023
- [Background] Kaynak BA, Tas S, Salkin Y. The accuracy and reliability of the Turkish version of the Fonseca anamnestic index in temporomandibular disorders. Cranio. 2023 Jan;41(1):78-83. doi: 10.1080/08869634.2020.1812808. Epub 2020 Aug 25. PMID 32840464
- [Background] Kim HS, Yun PY, Kim YK. A clinical evaluation of botulinum toxin-A injections in the temporomandibular disorder treatment. Maxillofac Plast Reconstr Surg. 2016 Jan 28;38(1):5. doi: 10.1186/s40902-016-0051-7. eCollection 2016 Dec. PMID 26855937
- [Background] Komino M, Shiga H. Changes in mandibular movement during chewing of different hardness foods. Odontology. 2017 Oct;105(4):418-425. doi: 10.1007/s10266-016-0292-z. Epub 2017 Feb 1. PMID 28150182
- [Background] Kwon KH, Shin KS, Yeon SH, Kwon DG. Application of botulinum toxin in maxillofacial field: part I. Bruxism and square jaw. Maxillofac Plast Reconstr Surg. 2019 Oct 1;41(1):38. doi: 10.1186/s40902-019-0218-0. eCollection 2019 Dec. PMID 31649901
- [Background] Lee CM, Huxley RR, Wildman RP, Woodward M. Indices of abdominal obesity are better discriminators of cardiovascular risk factors than BMI: a meta-analysis. J Clin Epidemiol. 2008 Jul;61(7):646-53. doi: 10.1016/j.jclinepi.2007.08.012. Epub 2008 Mar 21. PMID 18359190
- [Background] Lee WK, Bae JH, Hu KS, Kato T, Kim ST. Anatomical recommendations for safe botulinum toxin injection into temporalis muscle: a simplified reproducible approach. Surg Radiol Anat. 2017 Mar;39(3):263-269. doi: 10.1007/s00276-016-1739-1. Epub 2016 Sep 8. PMID 27631881
- [Background] Monteiro DR, Zuim PR, Pesqueira AA, Ribeiro Pdo P, Garcia AR. Relationship between anxiety and chronic orofacial pain of temporomandibular disorder in a group of university students. J Prosthodont Res. 2011 Jul;55(3):154-8. doi: 10.1016/j.jpor.2010.11.001. Epub 2010 Nov 26. PMID 21112271
- [Background] Mumcu G, Inanc N, Ergun T, Ikiz K, Gunes M, Islek U, Yavuz S, Sur H, Atalay T, Direskeneli H. Oral health related quality of life is affected by disease activity in Behcet's disease. Oral Dis. 2006 Mar;12(2):145-51. doi: 10.1111/j.1601-0825.2005.01173.x. PMID 16476035
- [Background] Nasri-Heir C, Epstein JB, Touger-Decker R, Benoliel R. What should we tell patients with painful temporomandibular disorders about what to eat? J Am Dent Assoc. 2016 Aug;147(8):667-71. doi: 10.1016/j.adaj.2016.04.016. Epub 2016 Jun 11. PMID 27301850
- [Background] Patel J, Cardoso JA, Mehta S. A systematic review of botulinum toxin in the management of patients with temporomandibular disorders and bruxism. Br Dent J. 2019 May;226(9):667-672. doi: 10.1038/s41415-019-0257-z. PMID 31076698
- [Background] Pedroni CR, De Oliveira AS, Guaratini MI. Prevalence study of signs and symptoms of temporomandibular disorders in university students. J Oral Rehabil. 2003 Mar;30(3):283-9. doi: 10.1046/j.1365-2842.2003.01010.x. PMID 12588501
- [Background] Reis JP, Macera CA, Araneta MR, Lindsay SP, Marshall SJ, Wingard DL. Comparison of overall obesity and body fat distribution in predicting risk of mortality. Obesity (Silver Spring). 2009 Jun;17(6):1232-9. doi: 10.1038/oby.2008.664. Epub 2009 Feb 5. PMID 19197258
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Tarkowska A, Katzer L, Ahlers MO. Assessment of masticatory performance by means of a color-changeable chewing gum. J Prosthodont Res. 2017 Jan;61(1):9-19. doi: 10.1016/j.jpor.2016.04.004. Epub 2016 May 17. PMID 27211494
- [Background] Torrance GW, Feeny D, Furlong W. Visual analog scales: do they have a role in the measurement of preferences for health states? Med Decis Making. 2001 Jul-Aug;21(4):329-34. doi: 10.1177/0272989X0102100408. PMID 11475389
- [Background] Villa S, Raoul G, Machuron F, Ferri J, Nicot R. Improvement in quality of life after botulinum toxin injection for temporomandibular disorder. J Stomatol Oral Maxillofac Surg. 2019 Feb;120(1):2-6. doi: 10.1016/j.jormas.2018.10.007. Epub 2018 Oct 29. PMID 30385428
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679